CLINICAL TRIAL: NCT02499952
Title: A Phase II Single-Arm Multi-Center Trial Evaluating the Efficacy of Pembrolizumab in the Treatment of Subjects With Incurable Platinum-Refractory Germ Cell Tumors: Hoosier Cancer Research Network GU14-206
Brief Title: Pembrolizumab in Subjects With Incurable Platinum-Refractory Germ Cell Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Efficacy
Sponsor: Nasser Hanna, M.D. (Other)
Collaborators: Hoosier Cancer Research Network (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Nasser Hanna, M.D., Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU14-206
Record Dates: First submitted 2015-07-08; First posted 2015-07-16 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Germ Cell Neoplasms; Testicular Neoplasms; Non Seminomatous Germ Cell Tumors; Mediastinal Neoplasms; Genital Neoplasms, Male; Genital Neoplasms, Female; Ovarian Neoplasms
Keywords: Pembrolizumab; MK-3475; PMNSGCT; PD-L1; Non Seminomatous Germ Cell Tumors
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Testicular Neoplasms; Nonseminomatous germ cell tumor; Mediastinal Neoplasms; Genital Neoplasms, Male; Genital Neoplasms, Female; Ovarian Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental Arm (Experimental): Pembrolizumab
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 200mg IV every 3 weeks until progressive disease, unacceptable toxicity, or after 52 weeks of therapy.
  Other Names: MK-3475

SUMMARY:
This is an open label, multi-institutional, single arm phase II trial of pembrolizumab in patients with incurable platinum refractory germ cell tumors. No randomization or blinding is involved.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

Eligible subjects must have received initial cisplatin-based combination therapy, such as bleomycin-etoposide-cisplatin (BEP), cisplatin-etoposide (EP), etoposide-ifosfamide-cisplatin (VIP), or similar regimens AND demonstrated progression following the administration of at least one 'salvage' regimen for advanced germ cell neoplasm, such as high dose chemotherapy, paclitaxel-ifosfamide-cisplatin (TIP), or vinblastine-ifosfamide-cisplatin (VeIP).

INVESTIGATIONAL TREATMENT:

Pembrolizumab 200mg IV every 3 weeks until progression or toxicity. Treatment will continue for up to 52 weeks in the absence of prohibitive toxicities or disease progression.

The following screening labs to demonstrate adequate organ function must be performed within 10 days of treatment initiation:

Hematological:

* Absolute neutrophil count (ANC) ≥1,500 /mcL
* Platelets ≥100,000 / mcL
* Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or hematopoietin (EPO) dependency (within 7 days of assessment)

Renal:

* Serum creatinine ≤1.5 X upper limit of normal (ULN) OR
* Measured or calculated creatinine clearance ≥60 mL/min for subject with creatinine levels >1.5 X institutional ULN
* Glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl)

Hepatic:

* Serum total bilirubin ≤ 1.5 X ULN OR
* Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
* Albumin >2.5 mg/dL

Coagulation:

* International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0 or 1 within 14 days prior to registration for protocol therapy.
* Subjects must have histological or serological proof of metastatic germ cell neoplasm (gonadal or extragonadal primary) with disease not amenable to cure with either surgery or chemotherapy. Subjects with seminoma and non-seminoma are eligible, as are women with ovarian GCTs.
* Subjects must have evidence of recurrent or metastatic carcinoma by one or more of the following: the appearance of metastatic disease on chest x-ray or CT scan, or the appearance of rising tumor marker: AFP or beta-HCG. NOTE: If a rising tumor marker is the only evidence of progressive disease, at least 2 consecutive rising values at least one week apart are needed. Subjects with only evidence of disease as rising tumor marker AFP and beta-HCG will be provided alternate causes of increased serum levels of these markers are not present, such as cross reaction with luteinizing hormone (LH) (that can be tested if needed by testosterone suppression of LH), hepatitis, use of marijuana, or second primary tumor, etc.
* Subjects must have received initial cisplatin based combination therapy, such as bleomycin-etoposide-cisplatin (BEP), cisplatin-etoposide (EP), etoposide-ifosfamide-cisplatin (VIP), or similar regimens AND demonstrated progression following the administration of at least one 'salvage' regimen for advanced germ cell neoplasm, such as high dose chemotherapy, paclitaxel-ifosfamide-cisplatin (TIP), or vinblastine-ifosfamide-cisplatin (VeIP).
* "Failure" of prior therapy is defined as: a >25% increase in the products of perpendicular diameters of measurable tumor masses during prior therapy which are not amenable to surgical resection; the presence of new tumors which are not amenable to surgical resection; an increase in AFP or beta-hCG (two separate determinations at least one week apart are required if rising tumor markers are the only evidence of failure). NOTE: Subjects with clinically growing "teratoma" (normal declining tumor markers and radiographic or clinical progression) should be considered for surgery.
* Subjects are eligible after first line platinum based chemotherapy if their disease has relapsed and they have Primary Mediastinal Non Seminomatous Germ Cell tumor (PMNSGCT) or late relapse (> 2 years) not amenable to surgical resection.
* Subjects must be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g., inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the sponsor investigator
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication . Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Measurable disease according to RECIST v1.1 obtained by imaging within 28 days prior to registration.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events (AE) due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. NOTE 1: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. NOTE 2: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e,. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Presence of interstitial lung disease or history of pneumonitis requiring treatment with corticosteroids.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with PD-1, PD-L1, or CTLA-4 inhibitors.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, M.D., Study Chair — Hoosier Cancer Research Network
Locations (2):
- United States (2):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adra N, Einhorn LH, Althouse SK, Ammakkanavar NR, Musapatika D, Albany C, Vaughn D, Hanna NH. Phase II trial of pembrolizumab in patients with platinum refractory germ-cell tumors: a Hoosier Cancer Research Network Study GU14-206. Ann Oncol. 2018 Jan 1;29(1):209-214. doi: 10.1093/annonc/mdx680. PMID 29045540
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Arm
Started | 12
Completed | 2
Not Completed | 10
Not completed — Lost to Follow-up | 1
Not completed — Death | 9

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Arm
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 38 [27 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Location Of Primary Tumor [Count of Participants; unit: Participants]
  Testis | 11
  Retroperitoneum | 0
  Mediastinum | 1
Tumor Histology [Count of Participants; unit: Participants]
  Seminoma | 0
  Nonseminoma | 12
Predominant Histology [Count of Participants; unit: Participants]
  Choriocarcinoma | 3
  Embryonal carcinoma | 5
  Teratoma | 1
  Yolk sac tumor | 3
Number of Previous Chemotherapy Regimens [Count of Participants; unit: Participants]
  1 | 1
  2 | 0
  3 | 7
  4 | 2
  5 | 1
  6 | 1
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead
  Participants
    ECOG 0 | 5
    ECOG 1 | 7
Metastatic Site(s) [Number; unit: participants] — The overall count of metastatic location(s). Subjects may have metastasis at multiple locations.
  participants
    Retroperitoneum | 5
    Pulmonary | 9
    Non Pulmonary Visceral Metastasis | 5

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR)
Description: CBR of single agent pembrolizumab in subjects with refractory germ cell tumors (GCTs), determined by sum of complete responses, partial responses, and stable disease for at least 3 months using Immune Related Response Criteria (irRC).
  Complete Response(irPR): Disappearance of all lesions in two consecutive observations not less than 4 wk apart.
  Partial Response (irPR): decrease in tumor burden ≥50 %relative to baseline confirmed by a consecutive assessment at least 4 wk after first documentation.
  Stable Disease (irSD): not meeting criteria for irCR or irPR, in absence of irPD.
Time Frame: up to 18 weeks
Measure: Number; unit: percentage of participants w/ clinical b
Arm/Group | Experimental Arm
Number analyzed (Participants) | 12
percentage of participants w/ clinical b | 0

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability Using Common Terminology Criteria for Adverse Events (CTCAE) V4.
Description: Toxicity and tolerability of pembrolizumab in subjects with refractory GCTs. All grade 3 and higher adverse events are reported.
Time Frame: Every week while patient is receiving pembrolizumab, assessed for up to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 12
Participants
  Skin and subcutaneous tissue disorders | 1
  Noncardiac chest pain | 1
  Anemia | 1
  Sciatic pain | 1

3. Secondary Outcome: Disease Assessment for Overall Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) Criteria
Description: ORR of single agent pembrolizumab in subjects with refractory GCTs, determined by sum of complete responses and partial responses for at least 3 months using RECIST 1.1 criteria
Time Frame: From the start of treatment D1 every 6 weeks for initial 18 weeks, assessed for up to 52 weeks
Population: Data for this secondary outcome measure was not collected or analyzed due to the early termination of this study.
Arm/Group | Experimental Arm
Number analyzed (Participants) | 0

4. Secondary Outcome: Disease Assessment for Duration of Disease Response
Description: Duration of disease response
Time Frame: From the start of treatment D1 every 6 weeks for initial 18 weeks, assessed for up to 52 weeks
Population: Data for this secondary outcome measure was not collected or analyzed due to the early termination of this study.
Arm/Group | Experimental Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months.
Arm/Group | Experimental Arm
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=12)
ANEMIA (Blood and lymphatic system disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=12)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (4)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BLOOD AND LYMPHATIC SYSTEM DISORDERS (Blood and lymphatic system disorders) | 1 (1)
BLURRED VISION (Eye disorders) | 1 (1)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 3 (3)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
EDEMA LIMBS (General disorders) | 2 (2)
FATIGUE (General disorders) | 6 (8)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
FLU LIKE SYMPTOMS (General disorders) | 2 (2)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1)
LARYNGEAL HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER (Musculoskeletal and connective tissue disorders) | 2 (3)
NAUSEA (Gastrointestinal disorders) | 5 (5)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 1 (2)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1)
PHOTOPHOBIA (Eye disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 3 (4)
SKIN ATROPHY (Skin and subcutaneous tissue disorders) | 1 (2)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 4 (6)

LIMITATIONS AND CAVEATS:
This study was terminated early due to not meeting the primary efficacy endpoint at a pre-planned interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No